CLINICAL TRIAL: NCT07311629
Title: Perceived Safety and Security Against Workplace Violence Among Otolaryngology-Head and Neck Surgery Physicians: A Multicenter Cross-Sectional Survey Study in Turkey
Brief Title: Workplace Violence and Safety Perception Among ENT Physicians in Turkey
Status: Not yet recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sumeyra DOLUOGLU, Assoc. Prof. Sumeyra Doluoglu, MD Department of Otolaryngology - Head and Neck Surgery University of Health Sciences, Ankara Etlik City Hospital, Türkiye, Saglik Bilimleri Universitesi
Other Study IDs: Sumeyra Doluoglu; Sumeyra Doluoglu (Other: University of Health Sciences, Ankara Etlik City Hospital)
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Workplace Violence; Perceived Safety; Occupational Health; Otolaryngology-Head and Neck Surgery Physicians
Keywords: Workplace violence; Safety perception; Otolaryngology; Healthcare professionals; Turkey

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ENT Physicians: Otolaryngology-Head and Neck Surgery (ENT-HNS) specialist and resident physicians aged 18 years or older working in Turkey who voluntarily participate in the study.
  Interventions: Other: Online Survey Questionnaire

INTERVENTIONS:
Other: Online Survey Questionnaire — An anonymous, web-based questionnaire administered via Google Forms to assess demographic characteristics, workload, exposure to workplace violence, reporting behaviors, and perceived safety against workplace violence using a validated safety perception scale.

SUMMARY:
This multicenter, cross-sectional survey study aims to evaluate the perceived level of safety and security against workplace violence among otolaryngology-head and neck surgery (ENT-HNS) physicians in Turkey. The study investigates the association between exposure to workplace violence and perceived safety, as well as the adequacy of institutional support mechanisms. Data will be collected through an anonymous online questionnaire distributed nationwide. The findings are expected to contribute to awareness and the development of preventive strategies and institutional safety policies for healthcare professionals.

DETAILED DESCRIPTION:
Workplace violence against healthcare professionals represents a significant occupational hazard, particularly for physicians working in high-risk clinical settings. ENT-HNS physicians frequently encounter high patient volumes, emergency conditions, and invasive procedures, which may increase the risk of violent incidents.

This non-interventional, cross-sectional study will be conducted using an anonymous, online survey distributed to ENT-HNS specialists and residents across Turkey. The questionnaire includes demographic and professional characteristics, workload indicators, exposure to different types of workplace violence (verbal, physical, and threats), reporting behaviors, and perceived safety levels measured using the "Healthcare Professionals' Safety and Security Perception Scale Against Violence."

The study involves minimal risk, limited to possible psychological discomfort due to recalling prior experiences of violence. No identifying information will be collected, and all data will be stored securely. Results will be reported in aggregate form only.

ELIGIBILITY:
Inclusion Criteria:

* Licensed ENT-HNS specialist or resident physician
* Aged 18 years or older
* Willingness to participate and provide informed consent

Exclusion Criteria:

* Physicians from other medical specialties
* Surveys with more than 20% missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Otolaryngology-Head and Neck Surgery (ENT-HNS) specialist and resident physicians aged 18 years or older working in Turkey who voluntarily participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Safety Score Against Workplace Violence | At survey completion (single time point, baseline assessment)
  Total score obtained from the Healthcare Professionals' Safety and Security Perception Scale Against Violence, a self-administered questionnaire assessing perceived safety and security in the workplace.
  The scale consists of items scored on a Likert-type scale, with a minimum score of 0 and a maximum score of 10.
  Higher scores indicate a higher perceived level of safety and security against workplace violence.

SECONDARY OUTCOMES:
Number of Participants Reporting Exposure to Workplace Violence | At survey completion (single time point, baseline assessment)
  Self-reported exposure to workplace violence, categorized as verbal violence, physical violence, and threats, assessed using a structured questionnaire developed for this study.
Correlation Between Perceived Safety Score and Exposure to Workplace Violence | At survey completion (single time point, baseline assessment)
  Correlation between:
  Perceived Safety Score measured by the Healthcare Professionals' Safety and Security Perception Scale Against Violence (continuous total score, range 0-10), and
  Exposure to workplace violence (yes/no), assessed via self-reported questionnaire.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.
  De-identified data may be available from the corresponding investigator upon reasonable request, subject to ethics committee approval.